CLINICAL TRIAL: NCT06513351
Title: Logistic Regression Prediction Model vs. Standard of Care for Prediction of Postpartum Hemorrhage - A Pragmatic Randomized Controlled Trial
Brief Title: A Pragmatic Randomized Controlled Trial to Predict Postpartum Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holly Ende (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Holly Ende, Associate Professor of Anesthesiology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 240187
Record Dates: First submitted 2024-07-02; First posted 2024-07-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Post Partum Hemorrhage
Keywords: Post Partum Hemorrhage; Cesarean Section; Vaginal Birth; Risk Prediction
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Single Center Pragmatic Randomized Controlled Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care - Comparator Arm A (No Intervention): Standard Care, which includes a category-based risk assessment tool as part of nursing admission workflow. The prophylactic interventions in the intervention are recommended by the tool but not specifically tied to provider-facing clinical decision support.
- Novel PPH Risk Prediction Model - Comparator Arm B (Active Comparator): Standard Care with addition of a recently developed, novel PPH risk prediction model.
  Interventions: Behavioral: Novel PPH Risk Prediction Model - Comparator Arm B

INTERVENTIONS:
Behavioral: Novel PPH Risk Prediction Model - Comparator Arm B — Patients in this group will receive the standard care risk assessment with the addition of a recently developed, novel PPH risk prediction model, which will automatically calculate a patient's numerical risk of hemorrhage based on 21 risk factors. Elevated risk of hemorrhage (>=3% predicted risk), as predicted by the model, will be linked to clinical decision support, including a best practice advisory with recommendations presented to providers for consideration when they access the patient's electronic health record.
  Arms: Novel PPH Risk Prediction Model - Comparator Arm B

SUMMARY:
This research project aims to enhance the safety of childbirth by using advanced computer models to predict the risk of postpartum hemorrhage (PPH).

PPH is a significant concern for mothers during and after delivery. Current risk assessment tools are basic and do not adapt to changing conditions. This study will investigate whether a new and recently validated model for predicting PPH, combined with a provider-facing Best Practice Advisory (BPA) regarding currently recommended strategies triggered by an increased predicted risk, can improve perinatal outcomes.

This study will compare the current category based risk assessment tool with a new, enhanced prediction model which calculates risk based on 21 factors, automatically updates as new information becomes available during labor and, if elevated, provides a provider-facing Best Practice Advisory (BPA) recommending consideration of strategies that are institutionally agreed to represent high-quality practice.

Investigators hypothesize that the enhanced care approach will result in improved perinatal outcomes.

The goal of the study is to improve the wellbeing of mothers during childbirth by harnessing the power of modern technology and data analysis.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a common complication following vaginal or cesarean delivery and contributes significantly to maternal morbidity and mortality in the United States. There are numerous clinical factors which contribute to a patient's risk of developing PPH. Utilization of an evidence-based tool for PPH risk prediction is recommended by national societies and required by the Joint Commission.

Most currently used tools are category based and assign a low, medium, or high risk of hemorrhage. These tools fail to take advantage of the vast amounts of data and computing power available via modern electronic medical records. Predictive modeling and informatics-based solutions could help to modernize PPH risk prediction and improve patient outcomes.

This study proposes to continue standard of care risk assessment for all patients, including those randomized to the intervention arm (ARM B). Those patients in the intervention arm (ARM B) will have an additional risk prediction displayed, which will show the quantitative output from the logistic regression PPH risk prediction model, (validated in a previous study). In addition to this display, patients above a preset threshold of 3% risk will have a Best Practice Advisory (BPA) deployed to clinicians with recommended actions. These recommended actions, including the prophylactic use of tranexamic acid and second-line uterotonics, are supported by best evidence in those patients deemed to be at elevated a priori risk of PPH. These prophylactic treatments are accepted standard of care for those patients deemed high risk, and may be administered, at the discretion of the covering clinician, to patients rated high risk by the current risk assessment tool in the comparator arm (Arm A) of the study. The recommendations within the best practice advisory serve as a reminder of best practices as defined by the department and providers are not forced to follow the recommendations of the best practice advisory.

ELIGIBILITY:
Inclusion Criteria:

* All vaginal and cesarean deliveries occurring at Vanderbilt University Medical Center

Exclusion Criteria:

* All patients will be randomized at the time of admission to the obstetric service. Patients who are discharged prior to delivery will be excluded from subsequent analysis. Any patients with a pre-delivery planned hysterectomy (for placenta increta or percreta) will be excluded from the treatment algorithm and primary analysis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Numerical hierarchical composite score of postpartum morbidity and mortality at hospital discharge | Date of randomization to Postpartum hospital discharge (usually 2-4 days)
  Patients will be assigned the most severe morbidity and mortality outcome score based on a range of criteria from 1 to 7 with 1 being the least severe and 7 being the most severe outcome. 1 is Estimated blood loss <1000 mL, 2 is Estimated blood loss >=1000 mL, 3 is Mechanical treatment of hemorrhage (uterine tamponade device insertion, uterine compression suture), 4 is Post-delivery red blood cell transfusion, 5 is Uterine artery embolization, 6 is Hysterectomy due to bleeding, and 7 is Death.
  For example, a patient who experiences an estimated blood loss >=1000mL and does not experience another more serious outcome would receive a score of 2, whereas a patient who requires a hysterectomy due to bleeding might meet several of the criteria, but would receive a score of 6, as this is the most severe criteria they experience.
Numerical hierarchical composite score of postpartum morbidity and mortality at 30 days postpartum | 30 days postpartum
  Patients will be assigned the most severe morbidity and mortality outcome score based on a range of criteria from 1 to 7 with 1 being the least severe and 7 being the most severe outcome. 1 is Estimated blood loss <1000 mL, 2 is Estimated blood loss >=1000 mL, 3 is Mechanical treatment of hemorrhage (uterine tamponade device insertion, uterine compression suture), 4 is Post-delivery red blood cell transfusion, 5 is Uterine artery embolization, 6 is Hysterectomy due to bleeding, and 7 is Death.
  For example, a patient who experiences an estimated blood loss >=1000mL and does not experience another more serious outcome would receive a score of 2, whereas a patient who requires a hysterectomy due to bleeding might meet several of the criteria, but would receive a score of 6, as this is the most severe criteria they experience.

SECONDARY OUTCOMES:
Estimated blood loss <1000 mL | Date of randomization up to 30 days postpartum
  Number of patients with estimated blood loss <1000mL
Estimated blood loss >=1000 mL | Date of randomization up to 30 days postpartum
  Number of patients with estimated blood loss >=1000mL
Mechanical treatment of hemorrhage | Date of randomization up to 30 days postpartum
  Number of patients who required mechanical treatment of hemorrhage (uterine tamponade device insertion, uterine compression suture)
Post-delivery packed red blood cell transfusion | Date of randomization up to 30 days postpartum
  Number of patients who required post-delivery packed red blood cell transfusion
Uterine artery embolization | Date of randomization up to 30 days postpartum
  Number of patients who required uterine artery embolization
Hysterectomy due to bleeding | Date of randomization up to 30 days postpartum
  Number of patients requiring a hysterectomy due to bleeding
Death | Date of randomization up to 30 days postpartum
  Number of patients who died within 30 days postpartum
Medication to prevent bleeding | Date of randomization to Postpartum hospital discharge (usually 2-4 days)
  Number of patients who received medication to prevent bleeding
Estimated blood loss (mL) | Date of randomization to Postpartum hospital discharge (usually 2-4 days)
  median and interquartile range for all patients
Total packed red blood cells (units) | Date of randomization to Postpartum hospital discharge (usually 2-4 days)
  median and interquartile range for all patients
Postpartum hospital length of stay (hours) | Date of randomization to Postpartum hospital discharge (usually 2-4 days)
  median and interquartile range for all patients
Acute myocardial infarction | Date of randomization up to 30 days postpartum
  Number of patients who experienced an acute myocardial infarction
Aneurysm | Date of randomization up to 30 days postpartum
  Number of patients who experienced an aneurysm
Acute renal failure | Date of randomization up to 30 days postpartum
  Number of patients who experienced acute renal failure
Acute respiratory distress syndrome | Date of randomization up to 30 days postpartum
  Number of patients who experienced acute respiratory distress syndrome
Amniotic fluid embolism | Date of randomization up to 30 days postpartum
  Number of patients who experienced amniotic fluid embolism
Cardiac arrest/ventricular fibrillation | Date of randomization up to 30 days postpartum
  Number of patients who experienced cardiac arrest/ventricular fibrillation
Conversion of cardiac rhythm | Date of randomization up to 30 days postpartum
  Number of patients who required conversion of cardiac rhythm
Disseminated intravascular coagulation | Date of randomization up to 30 days postpartum
  Number of patients who experienced disseminated intravascular coagulation
Blood transfusion | Date of randomization up to 30 days postpartum
  Number of patients who required a blood transfusion
Eclampsia | Date of randomization up to 30 days postpartum
  Number of patients who experienced eclampsia
Heart failure/arrest during surgery or procedure | Date of randomization up to 30 days postpartum
  Number of patients who experienced heart failure/arrest during surgery or procedure
Puerperal cerebrovascular disorders | Date of randomization up to 30 days postpartum
  Number of patients who experienced puerperal cerebrovascular disorders
Pulmonary edema/acute heart failure | Date of randomization up to 30 days postpartum
  Number of patients who experienced pulmonary edema/acute heart failure
Severe anesthesia complications | Date of randomization up to 30 days postpartum
  Number of patients who experienced severe anesthesia complications
Sepsis | Date of randomization up to 30 days postpartum
  Number of patients who experienced sepsis
Shock | Date of randomization up to 30 days postpartum
  Number of patients who experienced shock
Sickle cell disease with crisis | Date of randomization up to 30 days postpartum
  Number of patients who experienced sickle cell disease with crisis
Air and thrombotic embolism | Date of randomization up to 30 days postpartum
  Number of patients who experienced air and thrombotic embolism
Hysterectomy | Date of randomization up to 30 days postpartum
  Number of patients who required a hysterectomy
Temporary tracheostomy | Date of randomization up to 30 days postpartum
  Number of patients who required a temporary tracheostomy
Ventilation | Date of randomization up to 30 days postpartum
  Number of patients who required ventilation
Post-delivery ICU admission | Date of randomization up to 30 days postpartum
  Number of patients who required ICU admission following delivery
Time from delivery to OR for patients requiring operative repair | Date of randomization to Postpartum hospital discharge (usually 2-4 days)
  Time from delivery to entry into the operating room for dilation and curettage, or operative repair of vaginal/cervical laceration
Fetal APGAR score at 1 minute | 1 minute post-delivery
  The median and interquartile range of the APGAR score will be reported for all patients. The Apgar score is a method to quickly summarize the health of newborn children. The Apgar score is determined by evaluating the newborn baby on five simple criteria: appearance (skin color), pulse (heart rate), grimace (reflex irritability), activity (muscle tone) and respiration on a scale from 0 to 2. Apgar total score (obtained by summing up values from all five items) ranges from 0 to 10 with a score of 0 expressing the worst neonatal status and a score of 10 the best status.
Fetal APGAR score at 5 minutes | 5 minutes post-delivery
  The median and interquartile range of the APGAR score will be reported for all patients. The Apgar score is a method to quickly summarize the health of newborn children. The Apgar score is determined by evaluating the newborn baby on five simple criteria: appearance (skin color), pulse (heart rate), grimace (reflex irritability), activity (muscle tone) and respiration on a scale from 0 to 2. Apgar total score (obtained by summing up values from all five items) ranges from 0 to 10 with a score of 0 expressing the worst neonatal status and a score of 10 the best status.
Fetal APGAR score at 10 minutes | 10 minutes post-delivery
  The median and interquartile range of the APGAR score will be reported for all patients. The Apgar score is a method to quickly summarize the health of newborn children. The Apgar score is determined by evaluating the newborn baby on five simple criteria: appearance (skin color), pulse (heart rate), grimace (reflex irritability), activity (muscle tone) and respiration on a scale from 0 to 2. Apgar total score (obtained by summing up values from all five items) ranges from 0 to 10 with a score of 0 expressing the worst neonatal status and a score of 10 the best status.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Ende, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No